CLINICAL TRIAL: NCT07293052
Title: Comparison of Outcome Between Grisotti Flap Versus Reverse Mirror Grisotti Flap for Central Quadrant Breast Tumors
Acronym: GRISOTTI FLAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Hospital Lahore (Other)
Responsible Party: Principal Investigator, Aqeela Shirazi, Dr., Mayo Hospital Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MayoLahore
Record Dates: First submitted 2025-11-26; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Reconstruction
Keywords: Central Quadrant Breast; Grisotti flap; Reverse Mirror Grisotti Flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grisotti Flap (Experimental): Grisotti flap will be used in this arm for the oncoplastic breast surgery.
  Interventions: Procedure: Grisotti Flap
- Reverse Mirror Grisotti flap (Active Comparator): Reverse Mirror Grisotti flap will be used in this group for the oncoplastic breast surgery.
  Interventions: Procedure: Reverse Mirror Grisotti Flap

INTERVENTIONS:
Procedure: Grisotti Flap — The Grisotti flap is a local rotational flap used to reconstruct defects after removing a central breast cancer, often involving the nipple-areola complex (NAC). It uses tissue from the inferior pole of the breast to fill the central defect. The dermoglandular flap will be raised on infero-lateral perforators of intercostal arteries and will be rotated and advanced to fill the gap .
  Arms: Grisotti Flap
Procedure: Reverse Mirror Grisotti Flap — The reverse-mirror version is a modification where the flap is flipped and reoriented, using the internal mammary vessels as the primary blood supply. The dermoglandular flap will be raised on the medial perforators of internal mammary artery and will be rotated and advanced to fill the defect.
  Arms: Reverse Mirror Grisotti flap

SUMMARY:
Breast conservation surgery is equivalent to mastectomy for early stage breast cancer patients. Central quadrant tumours can be treated with various oncoplastic techniques with a satisfactory aesthetic outcome and low morbidity. Grisotti flap and reverse mirror grisotti flap are the favourable viable surgical options for central quadrant breast tumours. our hypothesis is that there is a difference in the outcome between Grisotti versus Reverse Mirror Grisotti flap in centrally located breast cancers.

DETAILED DESCRIPTION:
Breast cancer amongst women is the most common cancer and the second leading cause of deaths related to cancer worldwide.6 Its incidence is rising by 1% annually during 2012-2021, largely confined to localized-stage and hormone receptor-positive disease.1 A steeper increase in women < 50 years (1.4% annual) versus >50 years (0.7%) overall was significant only among White women. African/Pacific Islander women had the fastest increase in both age groups (2.7% for women <50 years and 2.5% for women > 50 years per year)1. Hence, young Asian ,American/Pacific Islander women had the second lowest rate in 2000 (57.4 per 100,000) but the highest rate in 2021 (86.3 per 100,000). 1 In a multitude of developed and emerging countries, including Pakistan, breast cancer is a cause of significant morbidity and mortality.1,2 The average age of developing a breast cancer among white American women is 61 years, however the average age for Pakistani women is 51.4 years.2 In the past, mastectomy was treatment of choice for any stage of breast cancer.9 However newer advancements resulting in early diagnosis, providing advancved systemic therapies and easy availability of radiotherapy facilities have paved the paths for breast conservations.7,9 Sometimes the size and location of the tumor leads to undesired aesthetic results which can be encountered when attempting resections with safe margins. The major part of the aesthetic problem after breast conservation surgery is due to large glandular defects and scars contractures.15 This is where oncoplastic techniques are used for the repair of resulting glandular defects without compromising the oncological outcomes.7,9,15 Breast oncoplastic surgery, integrating oncologic and plastic surgery principles, is increasingly prevailing in developed as well as developing countries. The technique involves precise and thorough planning of incisions,excisions, glandular reshaping and nipple areolar complex (NAC) repositioning for improved and symmetrical aesthetic outcomes.3 Oncoplastic breast surgery has hence become the standard of care in breast cancer owing to its feasibility,advances and oncological safety .5 Among the different quadrant tumours, centrally located breast tumours (CLBT) account for about 5-20% of all breast cancer cases.7,9 Because of their location CLBT pose special oncological and aesthetic concerns. Selecting an optimal surgical approach for CLBT remains debated till date, reflecting the complexity of balancing oncologic principles with aesthetic outcomes and local control.3 The resection of NAC is almost always necessary in central quadrant tumours and aesthetic outcomes are mostly poor if only a standard breast conservative therapy is performed.14 Oncoplastic approaches for centrally located breast tumours may include Grisotti flap, reverse mirror grisotti flap, latissimus dorsi flap, inferior pedicle flap, Melon slice, and round block techniques16. For centrally located breast tumours Grisotti flap technique has a short learning curve, quick to perform, with a low complication rate, satisfactory cosmetic outcome and no loss of body image in the post-operative period making it a more physiological procedure.7,13 The oncologic outcome of oncoplastic breast conservation was shown to be comparable to the classical mastectomy in cases of central breast tumors 10. The Grisotti technique consists of excising central quadrant breast tumor alongwith nipple areolar complex and mobilizing a dermo-glandular flap which is de-epithelized, rotated and advanced based on inferior and lateral pedicle in order to fill the glandular defect and reshape the breast, recreating a neo-areola.8,9 Grisotti flap is a partial mastectomy and an immediate volume replacement technique10 The Grisotti flap technique demonstrated superior patient satisfaction alongwith aesthetic and psycho-social outcomes while maintaining oncological safety that is comparable to that of mastectomy.Hence Grisotti flap technique is a standard alternative to mastectomy, particularly in patients prioritizing aesthetic outcomes. 4,6 Advances in oncoplastics have devised the modification of this original technique which involves the utilizing other vascular pedicles for the dermoglandular advancement and rotation.9 A reverse-mirror Grisotti flap, also known as a Reverse-Bay of Bengal modification, is a variation of the Grisotti flap technique used in breast cancer surgery. It is designed to reconstruct defects in the central breast quadrant after a breast conservation surgery. This modification involves re-orienting the flap medially where it is dependent mainly on the perforators of internal mammary artery for blood supply, potentially offering better aesthetic results and more versatile and robust blood supply. The Grisotti flap, despite its well known utility, has limitations, particularly in patients with non-ptotic breasts, where it may lead to fullness laterally and suboptimal cosmesis, the Reverse Bay of Bengal modification of the Grisotti flap is designed to address these limitations by preserving chest wall perforators and avoiding excessive lateral buldging.11 This technique hence offers a more cosmetic alternative for patients with central quadrant tumors requiring nipple-areola complex (NAC) excision.11

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed cases of breast cancer patients
2. Gender: Females
3. Age: 25-70 years
4. T1 (<2cm) and T2 (2-5cm) tumors with or without prior systemic therapy
5. Tumor located in the NAC or located within 2 cm of the edge of the areola

Exclusion Criteria:

1. Metastatic breast cancer
2. Inflammatory breast cancer
3. Patients not willing for post-operative radiotherapy
4. High tumour-breast ratio

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 106 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Flap viability | 7 days
  Absence of necrosis of new areola formed as seen clinically at 48 hours and 7th day postoperatively.
  Flap viability categories:
  A (None): No necrosis. B (Color Change): Color change suggesting impaired perfusion or ischemic injury.
  C (Partial Thickness): Partial thickness skin flap necrosis resulting in wound breakdown.
  D (Full Thickness): Full thickness skin flap necrosis.

SECONDARY OUTCOMES:
Cosmetic outcome | 7 days
  Cosmetic outcome will be explained with VAS (visual analogue scale) by the patient. The scale will range from 0-10 with 0 being categorized as worst cosmetic outcome and 10 being categorized as best cosmetic outcome.
Seroma formation | 7 days
  Seroma formation is the visible swelling at the operative site which will be confirmed and quantified by ultrasound on 7th post operative day with volume more than 20ml.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Informed consent will be obtained from all individual participants with diagnosis of central quadrant breast tumors as per operational definition, and data will be collected on predesigned proforma. Information will include name, age, gender, medical registration number, contact and residence.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: IPD could be provided after contacting with the principal investigator. Other researchers requiring information excluding personal data will be provided only for ethical and educational purposes.

REFERENCES:
- [Result] Abdelkader AA, El-Fayoumi T, Roushdy A, Asal MF. Comparison between conventional and oncoplastic breast surgeries regarding resection margins and local recurrences in breast cancer: Retrospective study. The Egyptian Journal of Surgery. 2023; 7;42(4).
- [Result] Ozgul H, Celik O, Sakar B, Celik A, Oener OZ. Postoperative patient satisfaction and oncological Outcomes of Grisotti flap vs. Total mastectomy: A retrospective analysis
- [Result] Koppiker CB, Noor AU, Joshi S, Mishra R, Sivadasan P, Sheikh S., et al.Pushing the Boundaries for Centrally Located Breast Tumors in Oncoplastic Breast Surgery: A Single Centre Audit. medRxiv. 2024 ; 25:2024-11.
- [Result] Siddiqui R, Alsuwaidi SA, Irkorucu O, Mehmood MH, Khan NA. The Increasing Importance of Breast Cancer in the United Arab Emirates. Asia Pac J Clin Oncol. 2025 Nov 15. doi: 10.1111/ajco.70050. Online ahead of print. PMID 41241761
- [Result] Giaquinto AN, Sung H, Newman LA, Freedman RA, Smith RA, Star J, Jemal A, Siegel RL. Breast cancer statistics 2024. CA Cancer J Clin. 2024 Nov-Dec;74(6):477-495. doi: 10.3322/caac.21863. Epub 2024 Oct 1. PMID 39352042
- Available data/document: Study Protocol — https://pdf.ac/0wrnmMTIc3

DOCUMENTS (1):
  • Study Protocol (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT07293052/Prot_000.pdf